CLINICAL TRIAL: NCT03800563
Title: The Safety and Efficacy of Laser Assisted Liposuction and Facial Autologous Fat Grafting With the LipoLife System
Brief Title: Laser Assisted Liposuction and Facial Autologous Fat Grafting With the LipoLife System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alma Lasers (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALM-Lipo-002
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2022-10-25 (Actual); Last update posted 2022-10-25 (Actual); Status verified 2019-11

CONDITIONS: Laser Assisted Liposuction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Laser assisted liposuction (Experimental): Laser Assisted Liposuction with the LipoLife system. Each subject underwent laser assisted liposuction surgery w/wo facial fat grafting , using the LipoLifeTM system. Pre-surgery evaluation visit was carried out 1 week prior to the surgery. Follow up visits to evaluate safety and efficacy will take place at 1, 3 and 6 months after the surgery.
  Interventions: Device: LipoLife system

INTERVENTIONS:
Device: LipoLife system — Abdominal/ Outer thighs Laser Assisted Liposuction. Five to twenty subjects out of the study group will also undergo facial fat grafting.

SUMMARY:
Multi-center, prospective, open-label, single arm study. The study aims to evaluate the safety and efficacy of Laser Assisted Liposuction procedure performed with the LipoLife system. The study will include twenty (20) eligible subjects, that are willing to undergo abdominal or outer thighs laser-assisted liposuction. Five to twenty (5-20) subjects out of this study group should also be eligible for facial fat grafting. Follow up visits to evaluate study endpoints will take place at 1, 3 and 6 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with excessive fat in the lower abdomen or subjects with excessive fat in the outer thighs that are willing to undergo laser-assisted liposuction
* Estimated fat harvesting of 1-3 liters
* Subjects (5-20) eligible for facial fat grafting of at least 5 cc for each cheek
* Between 18 and 70 years of age
* Provided written Informed Consent

Exclusion Criteria:

* Body Mass Index (BMI) >35
* Sever skin laxity
* Positive pregnancy test
* Current smoker
* Presence of known malignancy
* Active infection in the treatment area
* History of autoimmune disorder (e.g., Systemic Lupus Erythematosus [SLE])
* History of connective, metabolic or atrophic skin disease
* History of keloid scarring
* Chronic use (>7 consecutive days) of anticoagulants (such as aspirin) or NSAIDs within 15 days prior to enrollment
* Subjects with immune system diseases
* Subject unable to follow post-treatment instructions
* Any other reason that in the opinion of the investigator, prevents the subject from participating in the study or compromise the subject safety.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-11-06 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2020-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason N. Pozner, M.D., Principal Investigator — Sanctuary Plastic Surgery; Lior Heller, M.D., Principal Investigator — Yitzhak Shamir Medical Center
Locations (2):
- Sanctuary Plastic Surgery, Boca Raton, Florida, United States
- Yitzhak Shamir Medical Center, Be’er Ya‘aqov, Israel

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser Assisted Liposuction of Abdominal Excessive Fat: Laser Assisted Liposuction with the LipoLife system. LipoLife system: Abdominal/ Outer thighs Laser Assisted Liposuction. Added: "Each subject underwent laser assisted liposuction surgery w/wo facial fat grafting , using the LipoLifeTM system. Pre-surgery evaluation visit was carried out 1 week prior to the surgery. Follow up visits to evaluate safety and efficacy will take place at 1, 3 and 6 months after the surgery." Seven subjects out of the study group underwent facial fat grafting.
Period: Overall Study
Arm/Group | Laser Assisted Liposuction of Abdominal Excessive Fat
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Laser Assisted Liposuction: Laser Assisted Liposuction with the LipoLife system.
  LipoLife system: Abdominal/ Outer thighs Laser Assisted Liposuction. Seven subjects out of the study group underwent facial fat grafting.
Arm/Group | Laser Assisted Liposuction
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
  Israel | 15

OUTCOME MEASURES:

1. Primary Outcome: Correct Identification of Before and After Photographs
Description: Over 90% success in correct identification of before and after body contouring photos by blinded evaluators.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Laser Assisted Liposuction
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Time Frame: Duration of each subject's participation was up to 8 months from enrollment to termination. Adverse events data was to be reported at any time during or after the use of the study device.
Description: Definitions of adverse event and serious adverse event used to collect adverse event information do not differ from the clinicaltrials.gov Definitions
Groups:
- Laser Assisted Liposuction: Laser Assisted Liposuction with the LipoLife system.
  LipoLife system: Abdominal/ Outer thighs Laser Assisted Liposuction. Five to twenty subjects out of the study group will also undergo facial fat grafting.
Arm/Group | Laser Assisted Liposuction
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 2/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Laser Assisted Liposuction (N=20)
Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) — localized bleeding outside of skin blood vessels.
urinary track infection (Infections and infestations) | 1 (1) — An infection in the urinary system that begins when microorganisms cling to the opening of the urethra (the canal from the bladder) and begin to multiply.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03800563/Prot_SAP_001.pdf
  • Informed Consent Form (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT03800563/ICF_002.pdf